CLINICAL TRIAL: NCT02504203
Title: Can Earlier BCG Vaccination Reduce Early Infant Mortality? A Randomised Trial
Acronym: BCGR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to fewer than expected children enrolled and lower than expected overall mortality rate.
Sponsor: Bandim Health Project (Other)
Collaborators: Research Center for Vitamins and Vaccines, Statens Serum Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCG150501
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Infant Mortality; BCG
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: BCG and OPV at home visits (Active Comparator): Infants randomised to receive vaccines at home visits shortly after birth will receive one 0.05 ml dose of Mycobacterium bovis BCG live attenuated vaccine (BCG-Denmark 1331 (Statens Serum Institute) or BCG Japan (Japan BCG Laboratory) by intradermal injection in the left deltoid region. Dependent on national supply, infants will receive oral polio vaccine (OPV) at the time of BCG vaccination. For all children, the nurse will perform umbilical cord and skin care, encourage skin-to-skin contact to keep the new-born warm, examine and weigh the child at a home visit shortly after birth.
  Interventions: Biological: BCG-Denmark 1331 (Statens Serum Institute)
- Control: No vaccines at home visits (No Intervention): For all children, the nurse will perform umbilical cord and skin care, encourage skin-to-skin contact to keep the new-born warm, examine and weigh the child at a home visit shortly after birth. No vaccines will be administered at these home visits for children in the control arm.

INTERVENTIONS:
Biological: BCG-Denmark 1331 (Statens Serum Institute) — See above
  Other Names: BCG-Japan (Japan BCG Laboratory)
  Arms: Intervention: BCG and OPV at home visits

SUMMARY:
The purpose of this study is to determine whether BCG vaccination shortly after birth can reduce early infant mortality in a rural and an urban setting.

DETAILED DESCRIPTION:
Background: BCG and oral polio vaccines (OPV) at birth are associated with beneficial non-specific effects, reducing neonatal mortality by more than what can be explained by prevention of the target diseases. BCG is recommended at birth, but is often given much later, especially in rural areas. In two RCTs in Guinea-Bissau, BCG-at-birth reduced neonatal mortality in low birthweight (<2500g; LBW) children by 48% (95%CI: 18-67%) and in children with a birthweight >2500g (NBW), OPV+BCG vs BCG was associated with a 32% (95%CI: 0-55%) lower mortality.

WHO recommends home visits shortly after birth to reduce mortality, but vaccinations are not normally provided. If the vaccines indeed have profound effects on innate immunity and neonatal mortality in both LBW and NBW children many lives could be saved if BCG and OPV was provided earlier. Urban and rural clusters are randomised to home visits with and without vaccinations. All children participating in the study will be offered routine vaccines at village visits by the BHP team in the rural area. In the urban area, BCG and OPV will be provided at follow-up visits if the child has not yet received the vaccines. Thereby the study will provide earlier vaccination for all children.

Hypothesis: BCG+OPV at birth provided at village visits shortly after birth will reduce early infant mortality by 40%.

Methods: The study will be conducted in Biombo, Oio and Cacheu in rural Guinea-Bissau and in six suburban districts in the capital of Guinea-Bissau. In Guinea-Bissau home visits are not yet implemented as part of the routine program. Pregnant women will be offered to participate in the study at the time of pregnancy registration, which is conducted as part of the routine registration in the rural and urban health and demographic surveillance systems, respectively. Community key informants or mothers will communicate information on births to the BHP study team, and a study nurse will visit every new-born child shortly after a CKI or mother calls, if possible on the same day. Clusters will be randomised to receive immediate vaccination of their children shortly after birth or at the first visit by the BHP team in the rural area and at 2-months follow-up visits in the urban area.

Statistical analyses: The primary analysis of early infant non-accidental mortality will be assessed on a PP analysis stratifying for factors used in the randomization (Region, pre-study mortality level (high/low)) and sex, thus allowing different baseline hazards for boys and girls. To account for clustering we will employ cluster-robust variance estimates.

For the primary outcome, we will use Cox proportional hazards models, stratified for the above mentioned factors and with age as underlying time-scale. Deaths due to accidents will be censored.

The effect of early vaccination will be assessed for the following secondary outcomes:

* Non-accidental hospital admission
* Severe morbidity (composite outcome of non-accidental mortality and non-accidental hospital admissions)
* Consultations
* Growth
* Mid-upper-arm circumference
* Weight-for-age z-score
* BCG scarring
* Cost-effectiveness of providing BCG and OPV at home visits

Based on previous data from the rural HDSS in the areas where the current study will be conducted, the expected proportion of events (deaths and hospitalisation) between day 1 and the next home visit or 60 days of age, whichever comes first is 2.4% (unpublished data). The proportion of events are expected to be at least as high in the urban area. A recent trial in Ghana indicated that three home visits during the first week of life to promote essential new-born care practices and to weigh and assess children for danger signs was associated with an 8% (-12 to 25%) reduction in neonatal mortality. Based on pre-trial mortality data from the same rural clusters, the design effect is measured to be 1.43 (ratio of square of the standard errors for the cluster-adjusted/unadjusted HRs). Thus, in order to obtain 80% power to detect a reduction in early infant severe morbidity if the true reduction of BCG and OPV provided at home visits is larger than 40%, at least 6666 children need to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

• All children registered during pregnancy will be eligible for the study provided they have not yet received BCG at the date of the home visit.

Exclusion Criteria:

* Children born outside the cluster, and returning more than 72 hours after the delivery
* Children that the nurse evaluates to die within the next 24 hours.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2332 (Actual)
Dates: Start 2015-11; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Non-accidental mortality | 60 days after birth
  Non-accidental mortality between the home visit and the next follow-up visit by BHP, when all unvaccinated children who are home will be offered BCG or the date of registering a non-trial vaccine or 60 days, whichever comes first.

SECONDARY OUTCOMES:
Non-accidental hospital admission | 60 days after birth
  Non-accidental hospital admission between the home visit and the next follow-up visit by BHP, when all unvaccinated children who are home will be offered BCG or the date of registering a non-trial vaccine or 60 days, whichever comes first.
Severe morbidity | 60 days after birth
  Composite outcome of non-accidental mortality and non-accidental hospital admissions
All-cause consultations | 60 days after birth
  All-cause out-patient consultation between the home visit and the next follow-up visit by BHP, when all unvaccinated children who are home will be offered BCG or the date of registering a non-trial vaccine or 60 days, whichever comes first.
Mid-upper-arm circumference | 60 days after birth
  Development in mid-upper-arm circumference measured using a TALC insertion tape between enrollment and first visit by the BHP team will be assessed.
Weight-for-age z-score | 60 days after birth
  Development in weight between enrollment and first visit by the BHP team will be assessed using WHO's weight-for-age z-score reference.
BCG scarring | 6 months after birth
  Development of a BCG vaccination scar (yes/no) will be assessed.
Cost-effectiveness analysis of providing BCG at home-visits | 60 days after birth
  A cost effectiveness analysis seeking to measure the cost per death averted using a societal perspective, contrasting the costs of vaccine provision in the present programme and an outreach system as tested in the trial. The costs/savings associated with different rates of consultations and admissions will also be taken into account.
Cause specific mortality | 60 days after birth
  For every death a verbal autopsy will be made

CONTACTS AND LOCATIONS:
Overall Officials: Sanne M Thysen, MD, PhD, Principal Investigator — Bandim Health Project; Ane B Fisker, MD,PhD, Principal Investigator — Bandim Health Project; Amabelia Rodrigues, PhD, Principal Investigator — Bandim Health Project; Christine S Benn, MD,PhD,DMSc, Study Director — Research Center for Vitamins and Vaccines; Peter Aaby, PhD,DMSc, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537
- [Background] Thysen SM, Byberg S, Pedersen M, Rodrigues A, Ravn H, Martins C, Benn CS, Aaby P, Fisker AB. BCG coverage and barriers to BCG vaccination in Guinea-Bissau: an observational study. BMC Public Health. 2014 Oct 4;14:1037. doi: 10.1186/1471-2458-14-1037. PMID 25282475
- [Derived] Thysen SM, da Silva Borges I, Martins J, Stjernholm AD, Hansen JS, da Silva LMV, Martins JSD, Jensen A, Rodrigues A, Aaby P, Stabell Benn C, Fisker AB. Can earlier BCG-Japan and OPV vaccination reduce early infant mortality? A cluster-randomised trial in Guinea-Bissau. BMJ Glob Health. 2024 Feb 12;9(2):e014044. doi: 10.1136/bmjgh-2023-014044. PMID 38350670
- [Derived] Thysen SM, Jensen AKG, Rodrigues A, Borges IDS, Aaby P, Benn C, Fisker A. Can earlier BCG vaccination reduce early infant mortality? Study protocol for a cluster randomised trial in Guinea-Bissau. BMJ Open. 2019 Sep 24;9(9):e025724. doi: 10.1136/bmjopen-2018-025724. PMID 31551370